CLINICAL TRIAL: NCT04506970
Title: Predicting Placental Pathologies by Ultrasound Imaging of the Human Placenta During Gestation
Brief Title: Predicting Placental Pathologies by Ultrasound Imaging
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mauro H. Schenone, Principal Investigator, Mayo Clinic
Other Study IDs: 20-000991
Record Dates: First submitted 2020-07-23; First posted 2020-08-10 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Intrauterine Growth Restriction; Villitis; IUGR
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intrauterine Growth Restriction: Pregnant women carrying a fetus identified with intrauterine growth restriction during the third trimester (>28 weeks gestation)
  Interventions: Diagnostic Test: Comprehensive Doppler Ultrasound of the Placenta; Other: Verasonics Ultrasound scanner (ultra-sensitive Doppler imaging)
- Normal pregnancy: Pregnant women identified with an uncomplicated pregnancy during the third trimester (>28 weeks), matched for fetal sex and gestational age with women enrolled in the IUGR group.
  Interventions: Diagnostic Test: Comprehensive Doppler Ultrasound of the Placenta; Other: Verasonics Ultrasound scanner (ultra-sensitive Doppler imaging)

INTERVENTIONS:
Diagnostic Test: Comprehensive Doppler Ultrasound of the Placenta — Ultrasound measures to be collected include uterine artery (UtA) and umbilical artery (UA), systolic/diastolic (S/D) ratio, resistance index (RI), pulsatility index (PI) and presence of early diastolic notch.
Other: Verasonics Ultrasound scanner (ultra-sensitive Doppler imaging) — In addition, a Verasonics ultrasound scanner will be used for ultra-sensitive Doppler imaging. Data will be collected on vessel density, periphery-to-center vessel density ratio (VDR) and microvessel morphology.

SUMMARY:
Intrauterine growth restriction (IUGR) is caused when the placenta cannot provide enough nutrients to allow normal growth of the fetus during pregnancy. It is unclear why IUGR happens, but an increase in inflammatory T cells in the placenta known as villitis of unknown etiology (VUE) is observed in many IUGR infants. The investigators aim to develop ultrasound methods for diagnosing VUE to understand it's role in IUGR.

DETAILED DESCRIPTION:
Intrauterine growth restriction (IUGR) occurs in 3-10% of all pregnancies and is associated with significant morbidity and mortality during pregnancy, after birth and throughout the child's lifespan. IUGR is caused by the inability of the placental vasculature to provide enough oxygen and nutrients to support the fetus; yet, the mechanisms leading to disruption of placental vasculature are unknown. The placenta of ~50% of IUGR fetuses are infiltrated with inflammatory cells, specifically maternal T cells, which destroy placental blood vessels that support the fetus. This infiltration of T cells is known as villitis of unknown etiology (VUE). The diagnosis of VUE is problematic because it occurs without clinical signs and symptoms of maternal (or fetal) distress and puts the fetus at significant risk of demise. Additionally, VUE commonly recurs in subsequent pregnancies putting future offspring at risk. Yet, the exact prevalence of VUE and its significance in IUGR pathogenesis and outcomes are poorly understood as VUE is only diagnosed after the infant is outside the womb. Therefore, the study aims to recognize risk factors and cellular mechanisms associated with VUE and develop methods for diagnosing and treating VUE in utero, in order to improve infant health.

ELIGIBILITY:
Inclusion Criteria for IUGR study cohort:

* Pregnancy > 28 weeks gestation
* Diagnosis of Intrauterine Growth Restriction (IUGR) before admission for labor and delivery
* Weight > 110 lbs (50 kg)
* Ability to understand and provide written informed consent

Inclusion Criteria for control cohort:

* Pregnancy > 28 weeks gestation
* No known pregnancy complications at prenatal obstetrical visit (+/- 1 week gestational age of matched subject in IUGR cohort)
* Weight > 110 lbs (50 kg)
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Known immunodeficiency or pregnancy complication (i.e. preeclampsia or gestational diabetes)
* Known autoimmune disease (e.g., rheumatoid arthritis or systemic lupus erythematosus) or chronic hypertension
* Chronic, active viral infections, including HIV-1/2, HTLV-1/2, Hepatitis B or C
* Solid organ or transplant recipient
* Current smokers (tobacco exposure within 30 days of registration)
* Conceptions from assisted reproductive technology (prior Clomid use is allowed)
* Multiple gestation
* Ruptured membranes
* Pregnancy <28 weeks gestation
* Not planning on delivering at Mayo Clinic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from women obtaining prenatal care in the obstetrics clinic at Mayo Clinic in Rochester, Minnesota. This study will consist of two cohorts: 1) women diagnosed with intrauterine growth restriction (IUGR) and 2) women having uncomplicated pregnancies. Forty women will be enrolled after being diagnosed with IUGR. Based on prior clinical data it is expected that 50% will have a VUE diagnosis. Another cohort of 20 women having uncomplicated pregnancies will also be enrolled, matched for fetal sex and gestational age at ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schenone, MD, Principal Investigator — Mayo Clinic; Elizabeth Ann L Enninga, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from September 2020 through March 2023
Period: Overall Study
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Started | 40 | 20
Completed (One participant was diagnosed with FGR and originally enrolled into the FGR group but was determined not to have FGR at their next clinical and research scan; therefore, this participant crossed over into the control group.) | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (5.2) | 30.8 (3.9) | 31.4 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 38 | 17 | 55
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 33 | 18 | 51
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60
Gravidity [Mean (Standard Deviation); unit: Pregnancies] | 2.7 (1.58) | 1.9 (1.33) | 2.4 (1.53)
Maternal BMI at ultrasound [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (5.62) | 28.3 (4.2) | 28.5 (5.16)
Smoking [Count of Participants; unit: Participants] — Smoking status collected at baseline. Potential risk factor for pregnancy.
  Participants | 2 | 0 | 2
Hypertension [Count of Participants; unit: Participants] | 9 | 4 | 13
Preeclampsia [Count of Participants; unit: Participants] | 3 | 2 | 5
Gestational Diabetes [Count of Participants; unit: Participants] | 8 | 1 | 9
Hypothyroidism [Count of Participants; unit: Participants] | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Uterine Artery Indices Completed
Description: Measured by Doppler and 3D microvessel imaging, used to calculate outcomes 3-5
Time Frame: Gestational age of 34-36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 40 | 20
Participants | 13 | 3

2. Primary Outcome: Number of Patients With Umbilical Artery Indices Completed
Description: Measured by Doppler and 3D microvessel imaging, used to calculate outcomes 3-5
Time Frame: Gestational Age of 34-36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 40 | 20
Participants | 29 | 8

3. Primary Outcome: Systolic(S)/Diastolic(D) Ratio
Description: S = Systolic peak (max velocity); Maximum velocity during contraction of the fetal heart.
  D = End-diastolic flow; Continuing forward flow in the umbilical artery during the relaxation phase of the heartbeat.
  S/D ratio = (systolic / diastolic ratio)
Time Frame: Gestational Age of 34-36 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 34 | 11
ratio | 2.8 (0.7) | 2.3 (0.4)

4. Primary Outcome: Resistance Index (RI)
Description: Resistance index (RI) = (systolic velocity - diastolic velocity / systolic velocity)
Time Frame: Gestational Age of 34-36 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 29 | 8
Ratio | 0.6 (0.7) | 0.6 (0.08)

5. Primary Outcome: Pulsatility Index (PI)
Description: Pulsatility index (PI) = (systolic velocity - diastolic velocity / mean velocity)
Time Frame: Gestational age of 34-36 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 13 | 3
Ratio | 1.0 (0.2) | 0.7 (0.0)

6. Primary Outcome: Number of Participants With Placental Pathology Indicating Chronic Villitis
Description: Using the Amsterdam criteria, following delivery, placentae will be histologically examined for placental villitis (presence of maternal T cells) and graded by severity. High grade involves greater than 10 villi while low grade affects fewer than 10 villi.
Time Frame: Gestational age up to 42 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 40 | 20
Participants | 8 | 7

7. Secondary Outcome: Gestational Age at Birth
Description: The gestational age in weeks of when the baby was delivered.
Time Frame: Gestational age up to 42 weeks
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 40 | 20
Weeks | 39.2 (1.3) | 38.1 (1.5)

8. Secondary Outcome: Preterm Labor
Description: Pregnancy that delivered prior to 37 weeks gestational age
Time Frame: Gestational age up to 37 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 40 | 20
Participants | 2 | 0

9. Secondary Outcome: Birth Weight of Infant
Description: Weight of infant at time of birth
Time Frame: Gestational age up to 42 weeks
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
Number analyzed (Participants) | 40 | 20
Grams | 2598 (457) | 3348.5 (444)

ADVERSE EVENTS:
Time Frame: From enrollment during the third trimester (> 28 weeks gestation) till the mother gives birth. Max reporting period is from Gestational age of 28 weeks to 42 weeks, a maximum of 14 weeks.
Arm/Group | Intrauterine Growth Restriction | Normal Pregnancy
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT04506970/Prot_SAP_000.pdf